CLINICAL TRIAL: NCT02565368
Title: A Randomized, Open-label, Single Dose, 2-way Crossover Study to Compare the Pharmacokinetic Characteristics of CKD-395 0.5/1000 mg in Healthy Male Volunteers
Brief Title: A Clinical Study to Compare the Pharmacokinetic Characteristics of CKD-395 0.5/1000 mg in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 158BE15008
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RT group (Experimental): R: Reference drug(Duvie Tab. 0.5mg, Glucophage XR Tab. 1000mg) 1T T: Test drug(CKD-395 0.5/1000mg) 1T
  Interventions: Drug: Duvie Tab. 0.5mg, Glucophage XR Tab. 1000mg; Drug: CKD-395 0.5/1000mg
- TR group (Experimental): T: Test drug(CKD-395 0.5/1000mg) 1T R: Reference drug(Duvie Tab. 0.5mg, Glucophage XR Tab. 1000mg) 1T
  Interventions: Drug: Duvie Tab. 0.5mg, Glucophage XR Tab. 1000mg; Drug: CKD-395 0.5/1000mg

INTERVENTIONS:
Drug: Duvie Tab. 0.5mg, Glucophage XR Tab. 1000mg — single oral administration
  Other Names: Lobeglitazone Sulfate 0.5mg, Metformin HCl 1000mg
Drug: CKD-395 0.5/1000mg — single oral administration

SUMMARY:
This study is a randomized, open-label, single dose, 2-way crossover study to compare the pharmacokinetic characteristics of CKD-395 0.5/1000 mg in healthy male volunteers.

DETAILED DESCRIPTION:
To healthy male subjects of twenty six(26), following treatments are administered dosing in each period fed condition(high fat meals) and wash-out period is a minimum of 7 days.

Treatment A(Reference Drug): DuvieTM Tab. 0.5mg 1T + Glicophage XR Tab. 1000mg 1T Treatment B(Test Drug): CKD-395 0.5/1000mg Tab. 1T Pharmacokinetic blood samples are collected up to 48hrs. Safety and pharmacokinetic are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy man older than 19 years at the time of screening.
2. BMI more than 17.5kg/m2 and less than 30.5kg/m2 and weight more than 55kg
3. Subject without congenital or chronic diseases and no psychotic symptoms or findings from the medical examination.
4. Suitable subject who is determined by laboratory tests such as hematology tests, blood chemistry, urinalysis test according to the characteristics of the drug and screening tests such as ECG test.
5. Subject who fully understand the clinical trials after in-depth explanation given prior to the clinical study, decided to join the clinical trials by their will and signed consent form which approved by Chonbuk National University Hospital IRB.
6. Subjects who are able to comply with all scheduled visits, laboratory tests and other procedures.

Exclusion Criteria:

1. Subjects who has a history of blood, kidneys, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological or allergic diseases that is clinically significant (Except untreated asymptomatic seasonal allergies at the time of administration)
2. Subjects who has a history of gastrointestinal disease or gastrointestinal surgery which can affect drug absorption.
3. Subjects who show AST or AST > 2 times upper limit of normal range.
4. Subjects who drink Alcohol > 210g/week within 6 months prior to the screening.
5. Subjects who take the medication involved in other clinical trials or bioequivalence tests within three months before the first dose medication characters.
6. Subjects who show Systolic Blood Pressure ≥ 140 mmHg or Diastolic Blood Pressure ≥ 90 mmHg at screening.
7. Subjects who have history of alcohol or drug abuse, within 1 year
8. Subjects who treated with metabolizing enzyme inducers or inhibitors such as barbitals within 30days prior to the first dosing.
9. Smoker ( ≥ 20cigarettes/day)
10. Subjects who takes ETC or OTC medicine within 10days before the first IP administration.
11. Subjects who do the whole blood donation within two months or component blood donation within 1month prior to the first dosing.
12. Subjects who can increase risk due to clinical test and administration of drugs or has Severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of test results.
13. Patients with hypersensitivity to lobeglitazone or any other thiazolidinediones ( Rosiglitazone, Rioglitazone) and to Metformin or any other biguanides
14. Patients with severe heart failure or congestive heart failure of needing drug therapy
15. Patients with liver disease
16. Patients with severe renal disease
17. Patients with diabetes mellitus with ketoacidosis, diabetes coma and prior
18. Patients before or after surgery, with severe infections, severe trauma
19. Subjects with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
20. Patients with renal disease or renal failure caused by cardiovascular collapse, acute myocardial infarction, sepsis (Serum creatinine ≥ 1.5mg/dL or abnormal creatinie clearance)
21. Patients who had a test to injecting radioactive iodine in vein
22. Patients with severe infections or severe traumatic whole body injuries
23. Patients with undernourishment condition or starvation state or hyposthenia or hypopituitarism, or hypoadrenalism
24. Patients with respiratory failure, or stomach disease
25. Subjects who is not able to intake high fat meals
26. Subjects who is not able to comply with guidelines described in the protocol.
27. Subjects who is determined by investigator's decision as unsuitable for clinical trial participation.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
AUClast of Lobeglitazon and metformin | Lobeglitazone: 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs / Metformin: 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 48hrs
Cmax of Lobeglitazon and metformin | Lobeglitazone: 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs / Metformin: 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 48hrs

SECONDARY OUTCOMES:
AUCinf of Lobeglitazon and metformin | Lobeglitazone: 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs / Metformin: 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 48hrs
Tmax of Lobeglitazon and metformin | Lobeglitazone: 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs / Metformin: 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 48hrs
t1/2 of Lobeglitazon and metformin | Lobeglitazone: 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs / Metformin: 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 48hrs
CL/F of Lobeglitazon and metformin | Lobeglitazone: 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs / Metformin: 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 48hrs
Vd/F of Lobeglitazon and metformin | Lobeglitazone: 0(Pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48hrs / Metformin: 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 48hrs

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea